CLINICAL TRIAL: NCT05062733
Title: Prospective Observational Study About SEBBIN Gluteal Implants
Brief Title: SEBBIN Round, Anatomical and Biconvex Gluteal Implants
Status: Recruiting | Type: Observational
Sponsor: Groupe SEBBIN (Industry)
Responsible Party: Sponsor
Other Study IDs: PEC 20-07-001
Record Dates: First submitted 2021-09-21; First posted 2021-09-30 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Complication; Prosthesis Durability
MeSH Terms: conditions — Prosthesis Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is part of the clinical evaluation of SEBBIN silicone gel-filled gluteal implants, included in the technical file of the device. The aim of the study is to gather additional data about the safety and effectiveness of the device.

ELIGIBILITY:
Inclusion Criteria:

* The patient is a man or a woman ≥ 18 years old at the time of inclusion.
* The patient is planned for a unilateral or bilateral gluteal implant placement with SEBBIN implants as per investigator decision
* The patient has been informed of the study, has read the patient informed consent and provided consent for the study in writing.

Exclusion Criteria:

* Patient implanted with silicone implants somewhere else in the body.
* Patient candidate for implantation with custom-designed implants.
* Participation in another interventional clinical study (participation into an observational study is permitted) with a medicinal product or a medical device in the 30 days prior to enrolment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: The intended target population for the gluteal Implants is women or men, who desire an increase in volume of the gluteal region for aesthetic or reconstruction reason.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-11-20 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2035-03 (Estimated)

PRIMARY OUTCOMES:
Complication rate | At 10 years of follow-up

CONTACTS AND LOCATIONS:
Locations (2):
- Istituto Estetico Italiano, Roma, Italy
- Medical Clinic "Essential Aesthetics", The Hague, Netherlands